CLINICAL TRIAL: NCT00029042
Title: A Randomized Double Blind Controlled Intra-Patient Dose Escalation Phase II Trial of Infliximab in Pediatric Patients With Refractory Juvenile Rheumatoid Arthritis
Brief Title: Infliximab to Treat Children With Juvenile Rheumatoid Arthritis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 020081; 02-AR-0081
Record Dates: First submitted 2002-01-04; First posted 2002-01-07 (Estimated); Last update posted 2008-08-27 (Estimated); Status verified 2008-08

CONDITIONS: Juvenile Rheumatoid Arthritis
Keywords: MRI; Inflammation; Joint Disability; Imaging; Biologic Therapy; Rheumatoid Arthritis; Juvenile Rheumatoid Arthritis; JRA; Children; Joints; Joint Inflammation
MeSH Terms: conditions — Arthritis, Juvenile; Inflammation; Arthritis, Rheumatoid; Arthritis | interventions — Infliximab

INTERVENTIONS:
Drug: Infliximab

SUMMARY:
This study will determine whether a stepwise increase of the drug infliximab (Remicade® (Registered Trademark)) controls juvenile rheumatoid arthritis more effectively than a fixed dose. It will look at the safety and effectiveness of increasing the dose to a maximum of 15mg/kg body weight per dose, examining the drug's effect on bone and cartilage, and whether it can improve abnormal growth, metabolism and hormones. Infliximab is approved for treating adults with rheumatoid arthritis and Crohn's disease.

Children between 4 and 17 years of age with active juvenile rheumatoid arthritis who do not respond adequately to standard therapy may be eligible for this study.

Participants will receive nine infusions of infliximab during this 62-week study. The drug is given intravenously (IV, into a vein) over 2 hours. The first three infusions will be at a dose of 5 mg/kg of body weight. Children who improve on this regimen will receive another 6 infusions at the same dose. Children who do not significantly improve on 5 mg/kg at the end of 6 weeks (the third infusion) may continue with phase 2 of the study, in which they will be randomly assigned to receive either: 1) 6 additional doses of the drug at 5 mg/kg per dose, or 2) a gradually increased dose to a maximum of 15 mg/kg. In addition, all children will continue to take methotrexate at the same dose as when they entered the study.

Participants will visit the NIH Clinical Center 12 times (about every 8 weeks) during the study for the following tests and procedures:

* History and physical examination, including a complete joint exam
* Puberty assessment - breast development in girls, testicle size in boys, and pubic hair
* Height and weight measurements

Children will have imaging studies (x-rays, MRI and Dexa scan) at the beginning and end of the study and will collect a 24-hour urine sample before each infliximab infusion.

Patients may elect to have an endocrine evaluation. This involves Clinical Center hospitalizations for 1-1/2 days on visits 1, 4 and 12. Small amounts of blood will be drawn every 20 minutes (through an indwelling catheter to avoid multiple needle sticks) for 8 hours while the child sleeps. The blood will be examined for the normal rhythm of growth hormone and other substances in the body and how they are affected by arthritis.

Participants will complete a questionnaire once a year for 2 years to provide information on their health status and any problems that might be related to the study drug.

DETAILED DESCRIPTION:
Infliximab, a murine chimeric monoclonal antibody targeted against TNF-alpha has recently been licensed for the treatment of adult patients with established rheumatoid arthritis (RA). A double blind placebo controlled trial in children with juvenile rheumatoid arthritis (JRA) using a single dose fixed infusion regimen is currently ongoing. This dose finding study is designed to determine whether a clinically guided intravenous (iv) infusion regimen allowing for intra-patient dose escalation is superior in achieving a 70% clinical response to fixed dose administration of infliximab in children with a polyarticular course of JRA. We will model the pharmacokinetic profile in both phases of the study. We plan to enroll a maximum of 48 patients to allow for 36 patients to be randomized into the two treatment arms. In the first phase of the study all patients will receive a fixed dose of 5mg/kg/dose for a total of 3 infusions over 6 weeks (weeks 0, 2, 6). In the second phase at week 14, patients who have not achieved a 70% improvement will be randomized at a 2:1 ratio to either receive intra-patient dose escalation capped at 15mg/kg/dose every 8 weeks or continue to receive 5mg/kg/dose every 8 weeks in a blinded fashion. After 6 additional IV doses, patients will again be evaluated clinically, radiographically and serologically for clinical response. Patients who achieved a 70% response by week 14 will be kept on 5mg/kg/dose every 8 weeks for the trial duration of 62 weeks, but will not be included in the primary endpoint analysis. We also plan to evaluate patients endocrinologically and metabolically to determine the effect of TNF blockade on these systems.

ELIGIBILITY:
INCLUSION CRITERIA:

Age: Patients must be less than 18 years of age and greater than or equal to 4 years of age.

Diagnosis of pauciarticular, polyarticular or systemic onset JRA according to the 'Criteria for the diagnosis of Juvenile Rheumatoid Arthritis' with evidence of active disease including all of the features within each category:

Pauciarticular JRA (if patients continue to develop a polyarticular course):

1. active synovitis involving at least 4 swollen joints
2. tenderness or pain on movement of greater than 4 involved joints

Polyarticular JRA:

1. active synovitis involving at least 4 swollen joints
2. tenderness or pain on movement of greater than 4 swollen joints
3. elevated acute phase reactants (ESR greater than 20mm/hr or CRP greater than 0.8mg/dl)

Systemic onset JRA (if patients develop a polyarticular course):

1. active synovitis involving at least 4 swollen joints
2. tenderness or pain on movement of greater than 4 swollen joints
3. elevated acute phase reactants (ESR greater than 20mm/hr or CRP greater than 0.8mg/dl)

Disease onset at age less than16 years.

Informed Consent: All parent(s) or their legal guardian(s) must sign a document of informed consent indicating their understanding of the investigational nature and the risks of this study before any protocol related studies are performed (this does not include routine laboratory tests or imaging studies required to establish eligibility). Pediatric patients will be included in all discussions in order to obtain verbal or written assent.

All patients enrolled must have an incomplete response to methotrexate at a dosage of at least 0.75 mg/kg/week or a maximum of 25 mg/week orally or subcutaneously for a minimum of 12 weeks.

No other disease modifying anti-rheumatic drugs will be allowed while on study. Patients on combination DMARD therapy will have all DMARDs (except methotrexate) withdrawn at least 2 weeks prior to trial initiation. Patients must be off etanercept for 4 weeks prior to enrolling in this study.

Stable doses of non-steroidal anti-inflammatory drugs including selective Cox-2 inhibitors. Patients enrolling should be on stable NSIAD doses for at least 2 weeks. If currently not on NSAIDs, patients must not have been using them for 2 weeks.

Stable dose of prednisone (or equivalent amount of any other corticosteroid) equal or less than 0.4 mg/kg/day for at least four weeks. If currently not on corticosteroids, patients must not have been using them for 4 weeks.

Subject has negative PPD.

If anergy control skin tests and PPD are negative, Infectious Disease (ID) will be consulted and if cleared by the ID the patient will be included into the study.

EXCLUSION CRITERIA:

Pregnant women and nursing mothers, sexually active men or women of childbearing potential not practicing birth control. (Sexually active subjects of childbearing or child-fathering potential must be willing to use an acceptable form of birth control, which includes oral contraceptives, barrier methods with spermicides, intrauterine devices (IUD's), medroxyprogesterone acetate (Depo-Provera), progestin implants or intrauterine system or surgical sterilization. All post-menarche females or females greater than or equal to 12 years must test negative on a urine pregnancy test. Sexually active males and females will be instructed to use condoms).

Patients with other rheumatic diseases that may confound the analysis including but not limited to Lyme disease, post streptococcal reactive arthritis, psoriatic arthritis, spondyloarthropathy, systemic lupus erythematosus, other infectious or reactive arthritis, or Reiter's syndrome.

Previous treatment with iv infliximab at doses greater than 3mg/kg/dose every 8 weeks.

Poor venous access.

Treatment with any monoclonal antibody in the past other than infliximab.

Allergy to murine-derived products.

Previous history or ongoing infection with tuberculosis or pneumocystis and patients with acute or chronic infections requiring anti-microbial therapy, serious viral infections (e.g. hepatitis, herpes zoster, CMV or HIV) or fungal infections or history of recurrent serious bacterial infections.

History of live vaccinations within the past 3 months.

Confounding medical illness that in the judgment of the investigators would pose added risk for study participants (e.g. chronic hepatic, hematologic, neurologic, renal, or pulmonary disease).

Past medical history or be currently diagnosed with any solid organ or hematologic malignancies including lymphoproliferative diseases and leukemias.

History of substance abuse within the past 5 years.

History of psychiatric illnesses that in the opinion of psychiatric consultants would pose added risk for study participants.

Pre-existing or recent onset of demyelinating disorders or type I diabetes.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 48
Dates: Start 2002-01; Study Completion 2005-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS), Bethesda, Maryland, United States